CLINICAL TRIAL: NCT02202928
Title: Phase 2 Study of Autologous Tumor Lysate-pulsed DC-CIK Cell in Colorectal Cancer After Surgery
Brief Title: Adoptive Cell Therapy Plus Chemotherapy and Radiation After Surgery in Treating Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Jingzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Colorectal Cancer
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer; Neoplasms; Intestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases
Keywords: Colorectal cancer; DC-CIK; Autologous tumor lysate
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Intestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases | interventions — Radiotherapy; Drug Therapy; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemo-radiotherapy (Sham Comparator): After accepting concurrent radiotherapy and chemotherapy according to NCCN guidelines, patients will just regularly follow up.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy
- DC-CIK (Experimental): After accepting concurrent radiotherapy and chemotherapy according to NCCN guidelines, patients will receive 3 cycles of autologous tumor lysate pulsed DC-CIK treatment.
  Interventions: Biological: DC-CIK; Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Biological: DC-CIK — 8×10^9 autologous tumor lysate pulsed DC-CIK cells for each infusion, IV (in the vein) for four cycles, each cycle received four infusions with a 1 day interval.
  Arms: DC-CIK
Radiation: Radiotherapy — 45~50 Gy in 25-28 fractions.
Drug: Chemotherapy — Oxaliplatin 85mg/m2 IV over 2 hours, day 1; Leucovorin 400mg/m2 IV over 2 hours, day 1; 5-FU 400mg/m2 IV bolus on day 1, then 1200mg/m2/day for 2 days IV continuous infusion; Repeat every 2 weeks.
  Other Names: FOLFOX

SUMMARY:
The purpose of this study is to evaluate the efficacy of autologous tumor lysate-pulsed dendritic and cytokine-induced killer cells (DC-CIK) for colorectal cancer (CRC).

DETAILED DESCRIPTION:
60 patients with stageⅠ~ Ⅲ CRC, who had received surgery and kept their tumor tissue, will be randomly divided into group A (receive DC-CIK treatment, chemotherapy and radiotherapy) or group B (just receive chemotherapy and radiotherapy), and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of autologous tumor lysate pulsed DC-CIK cells treatment (every 4 weeks) and 4 cycles chemo-radiotherapy. Patients in group B will receive only 4 cycles chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18~80 years old;
* Histologically confirmed with colorectal cancer at stage Ⅰ~Ⅲ;
* Patients who can accept curative operations;
* Patients who have a life expectancy of at least 3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1.

Exclusion Criteria:

* Hemoglobin<8.0 g/dL,Platelet count <75 x 10^9/L; ALT, AST, BUN and Cr more than normal limits on 3.0 times ;
* Known or suspected allergy to the investigational agent or any agent given in association with this trial;
* Pregnant or lactating patients;
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection;
* Patients who are suffering from serious autoimmune disease;
* History of organ allograft;
* Patients who had distant metastases;
* Patients who had active infection;
* Prior use of any anti-cancer treatment in 30 days;
* Now or recently will join another experimental clinical study ;
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Quality of life (QOL) | 3 Years
Phenotypic analysis of T cells | 1 year
  The number of CD3+ (or CD8+ or CD4+ or CD56+) T cell

CONTACTS AND LOCATIONS:
Overall Officials: Ke N Zhang, Professor, Principal Investigator — Jingzhou Central Hospital
Locations (1):
- Jingzhou Central Hospital Immunotherapy center, Jingzhou, Hubei, China